CLINICAL TRIAL: NCT00602147
Title: Genetic Analysis of Toxicity Associated With High-Dose Melphalan
Brief Title: Studying Common Genetic Mutations Related to Mucositis in Patients With Multiple Myeloma Receiving High-Dose Melphalan
Status: Terminated | Type: Observational
Why Stopped: The original PI on this study left VICC, thus study was closed.
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stephen Brandt, Professor of Medicine, Cell and Developmental Biology, and Cancer Biology, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC HEM 0750; VU-VICC-HEM-0750; VU-VICC-070644
Record Dates: First submitted 2008-01-22; First posted 2008-01-28 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Mucositis; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: mucositis; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Mucositis; Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample or cheek cells will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective sample: People who have been diagnosed with multiple myeloma and have received high-dose melphalan.
  Interventions: Other: laboratory biomarker analysis
- Prospective sample: People who have been diagnosed with multiple myeloma and will be receiving high-dose melphalan.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Blood or cheek cells wil be collected.

SUMMARY:
RATIONALE: Studying blood or mouthwash samples in the laboratory from patients receiving melphalan for cancer may help doctors learn more about changes that occur in DNA, identify biomarkers related to cancer, and help predict how patients will respond to treatment.

PURPOSE: This clinical trial is studying common genetic mutations related to mucositis in patients with multiple myeloma receiving high-dose melphalan.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether single nucleotide polymorphisms (SNPs) in genes that encode the melphalan transporters are associated with the development and/or severity of mucositis in patients with multiple myeloma receiving high-dose melphalan.
* To determine whether SNPs in genes that influence melphalan metabolism are associated with the development and/or severity of mucositis in these patients.

OUTLINE: This is a multicenter study.

Blood or mouthwash samples are collected and DNA isolated from these specimens is analyzed for single nucleotide polymorphisms (SNPs) in LAT1 or other candidate genes. Public databases (i.e., dbSNP and HapMap) are reviewed to select representative SNPs for genotype analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma
* Receiving treatment with high-dose melphalan for an autologous stem cell transplantation at any of these facilities:

  * Vanderbilt University Medical Center
  * Nashville Veteran's Administration Medical Center (VAMC)
  * Seattle VAMC
  * San Antonio VAMC

PATIENT CHARACTERISTICS:

* Not pregnant

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No palifermin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have been diagnosed with multiple myeloma and have received or will be receiving high-dose melphalan.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Association between single nucleotide polymorphisms (SNPs) in genes that encode the melphalan transporters and development and/or severity of mucositis | 4 weeks
Association between SNPs in genes that influence melphalan metabolism and development and/or severity of mucositis | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Brandt, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee